CLINICAL TRIAL: NCT00146952
Title: Evaluation of a Vibrotactile Sensory Aid Developed by the US Navy to Combat Pilot Disorientation as a Prosthesis in Patients With Postural Imbalance and Spatial Disorientation
Brief Title: Use of a Vibrotactile Sensory Prosthesis in Patients With Postural Imbalance and Spatial Disorientation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Collaborators: Medical Research Council (Other Government)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: DNMCA-PR1077
Record Dates: First submitted 2005-09-05; First posted 2005-09-07 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2005-09

CONDITIONS: Vestibular Diseases; Peripheral Neuropathies; Proprioceptive Disorders; Hemispatial Neglect
Keywords: Hemineglects
MeSH Terms: conditions — Vestibular Diseases; Peripheral Nervous System Diseases; Somatosensory Disorders; Perceptual Disorders

INTERVENTIONS:
Device: Vibrotactile feedback

SUMMARY:
The investigators propose to explore the hypothesis that vibrotactile channels for indicating spatial orientation can be exploited as a sensory prosthesis. The specific research applications will be used for guiding visual orientation, to provide alternative feedback to vision and vestibular signals for controlling balance, and for directional and lateralisation cueing in patients with neglect syndromes. The programme will study whether vibrotactile feedback improves performance and also if it speeds rehabilitation when used as an adjunct to conventional therapy.

ELIGIBILITY:
Inclusion Criteria:

* Sensory impairments
* Unsteadiness

Exclusion Criteria:

* High strokes

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-01; Study Completion 2007-12

PRIMARY OUTCOMES:
Mean time reaction to the perturbation with the feedback

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Gresty, Pr, Principal Investigator — Imperial College London; Adolfo M Bronstein, Pr, MD, Study Director — Imperial College London; Christopher Kennard, Pr, MD, Study Director — Imperial College London; Masud Husain, Dr, Study Director — Imperial College London
Locations (1):
- Charing Cross Hospital, London, United Kingdom

REFERENCES:
- See also: Related Info — http://www1.imperial.ac.uk/medicine/about/divisions/neuro/npmdepts/clinneuroscience/movandbal/otology/mbprosthesis/